CLINICAL TRIAL: NCT06750510
Title: Digital Universal Parenting Program for Positive Parenting Behaviors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Andre Sourander, Professor, University of Turku
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BePresent
Record Dates: First submitted 2024-08-29; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-08

CONDITIONS: Parenting
Keywords: Parent-Training; Parenting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Participants assigned to this condition will receive the 8-weeks intervention
  Interventions: Behavioral: Digitally Delivered Parent Training

INTERVENTIONS:
Behavioral: Digitally Delivered Parent Training — The intervention is a universal, digitally delivered parenting program, including 5 themes with recommended length of 1 week each. The total length of the intervention is 8 weeks. The program focuses on positive parenting, encouraging to develop parenting skills that strengthen their relationships and communication with their children.

SUMMARY:
The goal of this study is to evaluate use and feasibility of digitally-delivered universal parenting program, which aims to promote positive parenting among guardians with 3 years-old children.

DETAILED DESCRIPTION:
The study will use a single-arm study design.The participants will use the universal parenting program for 8-weeks.

The intervention is a digital parent training program which focuses on positive parenting and encouraging to develop parenting skills that strengthen the relationships and communication with their children. The topics includes for example reinforcing child´s positive behavior, reducing conflict situations and planning situations advanced, managing daily transitions, and being present to child. The program includes 5 themes with recommended length of 1 week each. Each theme includes theory material, videos, examples, video practices and exercises. The program is fully digital and provided in a dynamic, web-based format. SMS and email reminders will be sent regularly during the program.

Recruitment: All parents with a 3-year old child who is participating in annual health checkup in child health clinic are considered eligible to the study and are asked to participate if they fulfil inclusion criteria and do not meet the exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Guardians having a child aged 3 years participating to annual health checkup in child health clinic.
* At least one of the guardians is able to understand the languages that intervention is provided in

Exclusion Criteria:

* Inability to read Finnish, Swedish, or English, as these are the languages that the intervention is provided in.
* No internet access

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Child´s affective reactivity | From baseline to 8-weeks follow-up
  The Affective Reactivity Index (ARI-P)

SECONDARY OUTCOMES:
Behaviour of the child | From baseline to 8-weeks follow-up
  10 questions about child´s behavior, focusing especially for child´s hyperactivity and conduct problems.
Daily activities | From baseline up to 8-weeks
  A questionnaire adapted from the Barkley Home Situations Questionnaire, which asks the parent to rate whether the child's behavior causes problems during specified daily routines
Completion rates | From baseline up to 8-weeks
  Completion and non-completion of the intervention for eight-week period by using the data recorded of the intervention platform
Intervention satisfaction | 8-weeks follow-up
  Questions related to satisfaction toward the intervention and acknowledged support in specific areas of parenting provided in the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Andre Sourander, Professor, MD, Study Director — University of Turku
Locations (2):
- Finland (2):
  - Kaisa Mishina, Turku
  - Wellbeing service counties, Turku

IPD SHARING:
Plan to Share IPD: Undecided